CLINICAL TRIAL: NCT04006301
Title: A First-in-Human Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of JNJ-74699157 in Participants With Advanced Solid Tumors Harboring the KRAS G12C Mutation
Brief Title: First-in-Human Study of JNJ-74699157 in Participants With Tumors Harboring the KRAS G12C Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108652; 2019-000565-21 (EudraCT Number); 74699157STM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Neoplasms; Advanced Solid Tumors; Non-small Cell Lung Cancer; Colorectal Cancer
Keywords: KRAS G12C
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with advanced solid tumors harboring the kirsten rat sarcoma virus homolog (KRAS) glycine-to-cysteine (G12C) mutation will receive oral administration of JNJ-74699157. The dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET) until the recommended Phase 2 Dose (RP2D) has been identified.
  Interventions: Drug: JNJ-74699157
- Part 2: Dose Expansion (Experimental): Two groups of participants with either non-small cell lung cancer or other solid tumors harboring KRAS G12C mutation will receive JNJ-74699157 at RP2D determined in Part 1.
  Interventions: Drug: JNJ-74699157

INTERVENTIONS:
Drug: JNJ-74699157 — Participants will receive JNJ-74699157 orally.
  Other Names: ARS-3248

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of JNJ-74699157 in participants with advanced solid tumors harboring a kirsten rat sarcoma virus homolog (KRAS) glycine-to-cysteine (G12C) mutation (Part 1: Dose escalation) and to determine the safety and preliminary antitumor activity of JNJ-74699157 at the RP2D regimen in participants with advanced solid tumors harboring a KRAS G12C mutation (Part 2: Dose expansion).

DETAILED DESCRIPTION:
KRAS is one of the most frequently mutated genes in human cancer. KRAS mutations lead to activation of cellular signaling that promotes tumor growth, and KRAS may therefore be a candidate target for anticancer therapy. This study will evaluate JNJ-74699157, a potent and specific, orally bioavailable inhibitor of the glycine-to-cysteine (G12C) mutant KRAS protein, which is found in non-small cell lung cancers and other solid tumor types. This study will enroll participants with advanced solid tumors harboring the KRAS G12C mutation and will be conducted in 2 parts. Part 1 (Dose Escalation) will be carried out in sequential cohorts of single or multiple participants at doses assigned by the study evaluation team to determine the MTD and RP2D of JNJ-74699157. Participants in Part 2 (Dose Expansion) will receive JNJ-74699157 at the RP2D determined in Part 1 to determine the safety and preliminary antitumor activity of the RP2D. Key efficacy assessments include radiographic imaging evaluations, physical examination, and tumor markers. Safety evaluations will include monitoring of adverse events, vital signs, laboratory evaluations, cardiac monitoring and physical examination findings. The study consists of a screening phase, treatment phase, and a post-treatment follow-up phase. An end-of-treatment visit will occur within 30 days of the last dose of study drug or prior to the start of a subsequent anticancer therapy, whichever comes first. The study duration will be up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Kirsten rat sarcoma virus homolog (KRAS) glycine-to-cysteine (G12C) mutation in tumor tissue or blood
* Histological documentation of disease: Part 1: Histologically or cytologically confirmed solid tumor malignancy that is metastatic or unresectable, Part 2: (a) unresectable, locally advanced (Stage IIIB) or metastatic (Stage IV) non-small cell lung cancer (NSCLC), (b) Solid tumor malignancy other than NSCLC that is metastatic or unresectable
* Received or was ineligible for standard treatment options. For NSCLC: previously received a platinum-containing chemotherapy regimen and an anti- programmed death-ligand 1 (PD1/PDL1) antibody, unless participant refused or was ineligible to receive such therapy; and for colorectal cancer (CRC): previously received at least 2 prior lines of therapy, including a fluoropyrimidine, oxaliplatin, and irinotecan, unless participant refused or was ineligible to receive such therapy. For Participants in France only: NSCLC: Previously received a platinum-containing chemotherapy regimen and an anti-PD1/PDL1 antibody or was ineligible to receive such therapy. CRC: Previously received at least 2 prior lines of therapy, including a fluoropyrimidine, oxaliplatin, and irinotecan or was ineligible to receive such therapy
* Measurable or evaluable disease: Part 1: either measurable or evaluable disease, Part 2: At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1

Exclusion Criteria:

* Symptomatic brain metastases or known leptomeningeal disease; asymptomatic brain metastases are allowed if they have been treated, have been stable for greater than or equal to (>=) 4 weeks as documented by radiographic imaging, and do not require prolonged (greater than [>]14 days) systemic corticosteroid therapy. Participants who have had complete surgical resection of or received stereotactic radiosurgery to less than or equal to (<=) 3 metastatic lesions will be permitted to enroll in the study within 14 days of such treatment if they have recovered from treatment, are clinically stable, and do not require prolonged systemic corticosteroid therapy as noted above
* Prior treatment with an inhibitor specific to KRAS G12C
* Prior solid organ transplantation
* History of malignancy (other than the disease under study) within 2 years before the first administration of study drug. Exceptions include squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 2 years
* Inability to take an orally administered drug, or medical disorder or prior surgical resection that may affect the absorption of the study drug. Such conditions include, but are not limited to, malabsorption syndrome, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or resection of the stomach or small bowel. If any of these conditions exist, the investigator should discuss with the sponsor to determine participant eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 2 years
  DLTs are defined as certain non-hematologic and hematologic toxicities of Grade 3 or higher.
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) | Up to 4 years
  An AE is any untoward medical occurrence in a participant who received study drug without regard to causal relationship.
Part 1 and Part 2: Number of Participants with AE's by Severity | Up to 4 years
  Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life threatening consequences; Grade 5: Death.
Part 2: Overall Response Rate (ORR) | Up to 4 years
  ORR is defined as the percentage of participants who have a partial response (PR) or better response as per RECIST v.1.1. PR criteria in solid tumors (RECIST) is greater than or equal to (>=) 30 percent (%) decrease in the sum of the diameters of all index lesions compared with baseline in 2 observations at least 4 weeks apart, in absence of new lesions or unequivocal progression of non-index lesions.

SECONDARY OUTCOMES:
Part 1 and Part 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-74699157 | Up to 4 years
  Cmax is the maximum observed plasma concentration.
Part 1 and Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-74699157 | Up to 4 years
  Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Part 1 and 2: Area Under Plasma-concentration Time Curve from Time 0 to Time of Last Quantifiable Concentration (AUC [0-last]) | Up to 4 years
  AUC (0-last) is the area under the plasma concentration-time curve from time zero to last observed quantifiable concentration.
Part 1 and 2: Percentage of KRAS G12C Protein in Tumor Tissue Covalently Bound with JNJ-74699157 or its Metabolites | Up to 4 Years
  Percentage of kirsten rat sarcoma virus homolog (KRAS) glycine-to-cysteine (G12C) protein in tumor tissue covalently bound with JNJ-74699157 or its metabolites will be evaluated using mass spectroscopy.
Part 1: Overall Response Rate | Up to 4 years
  ORR is defined as the percentage of participants who have a PR or better response as per RECIST v.1.1. PR criteria in solid tumors (RECIST) is >=30 percent % decrease in the sum of the diameters of all index lesions compared with baseline in 2 observations at least 4 weeks apart, in absence of new lesions or unequivocal progression of non-index lesions.
Part 1 and Part 2: Duration of Response (DOR) | Up to 4 years
  DOR is defined as the duration from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease (PD), as defined in the RECIST v1.1, or death due to any cause, whichever occurs first. PD is assessed if the sum of the diameters has increased by >=20% and >=5 millimeter (mm) from nadir (including baseline if it is the smallest sum).
Change From Baseline in QTc Interval Based on the Fridericia Correction (QTcF) Method | Baseline up to 4 years
  Change from baseline in QTcF intervals will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- United States (4):
  - Florida Cancer Specialists, Sarasota, Florida
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
- France (3):
  - Centre Leon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Wang J, Martin-Romano P, Cassier P, Johnson M, Haura E, Lenox L, Guo Y, Bandyopadhyay N, Russell M, Shearin E, Lauring J, Dahan L. Phase I Study of JNJ-74699157 in Patients with Advanced Solid Tumors Harboring the KRAS G12C Mutation. Oncologist. 2022 Jul 5;27(7):536-e553. doi: 10.1093/oncolo/oyab080. PMID 35325211